CLINICAL TRIAL: NCT02558543
Title: Subcutaneous Injection of Autologous Adipose Tissue-derived Stromal Vascular Fraction Into the Fingers of Patients With Systemic Sclerosis : Controlled Clinical Trial With Efficacy Assessment
Brief Title: Subcutaneous Injection of Autologous Adipose Tissue-derived Stromal Vascular Fraction Into the Fingers of Patients With Systemic Sclerosis
Acronym: scleradec2
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014-003321-17
Record Dates: First submitted 2015-08-31; First posted 2015-09-24 (Estimated); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Scleroderma, Systemic
MeSH Terms: conditions — Scleroderma, Systemic | interventions — Ringer's Lactate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stromal Vascular Fraction (Active Comparator): The injection is made for the patients of the both groups in the sub-dermic plan on the side faces of fingers distal and proximal or 4 times 0,25ml by finger, all in all every finger will be injected of 1ml of diluted Stromal Vascular Fraction ( experimental group) , or placebo (ringer lactate) ( placebo group)
  Interventions: Drug: Stromal Vascular fraction
- Placebo (Placebo Comparator): The injection is made for the patients of the both groups in the sub-dermic plan on the side faces of fingers distal and proximal or 4 times 0,25ml by finger, all in all every finger will be injected of 1ml of diluted Stromal Vascular Fraction ( experimental group) , or placebo ( placebo group)
  Interventions: Drug: Ringer lactate

INTERVENTIONS:
Drug: Stromal Vascular fraction
  Arms: Stromal Vascular Fraction
Drug: Ringer lactate
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
Systemic sclerosis (SSc) is an auto-immune orphan disease mainly characterized by an alteration of the microvascular network, and by cutaneous and visceral fibrosis. Hands are frequently affected, as a consequence of ischemic phenomena and cutaneous fibrosis.

. The injection of adipose autologous tissue is a common practice in plastic surgery, and has been known for over a century. Adipose tissue, originally used to increase volume, is also characterized by trophic properties associated to stromal vascular fraction (SVF), which contain multipotent stem cells, capable of tissue repair. Interestingly, some SVF cells can be angiogenic and anti-inflammatory, which could improve damage seen with SSc.

A prior study (the SCLERADEC protocol: ClinicalTrials.gov NCT01813279) has already allowed the safety and tolerance at 6 months of the subcutaneous injection of SVF in the fingers of twelve patients to be proven.

The encouraging results have encouraged us to propose a trial which would bear on a higher number of patients and include a control group.

DETAILED DESCRIPTION:
Systemic sclerosis (SSc) is an auto-immune orphan disease mainly characterized by an alteration of the microvascular network, and by cutaneous and visceral fibrosis. Hands are frequently affected, as a consequence of ischemic phenomena and cutaneous fibrosis. As a result, patients suffer from everyday disability, with consequences on their occupational activities and social contact, sometimes severely altering their quality of life. To date, no anti-fibrosis treatment has proven effective; existing vasodilation treatments are unfortunately not very effective, and are associated with adverse effects or restrictions. It is consequently of utmost importance that an effective treatment for sclerodermic hands be developed. The injection of adipose autologous tissue is a common practice in plastic surgery, and has been known for over a century. Adipose tissue, originally used to increase volume, is also characterized by trophic properties associated to stromal vascular fraction (SVF), which contain multipotent stem cells, capable of tissue repair. Interestingly, some SVF cells can be angiogenic and anti-inflammatory, which could improve damage seen with SSc. The injection of SVF into the fingers would also make it possible to control the production of the extracellular matrix and to improve the balance between fibrosis and fibrolysis, resulting in an improvement of cutaneous sclerosis.

A prior study (the SCLERADEC protocol: ClinicalTrials.gov NCT01813279) has already allowed the safety and tolerance at 6 months of the subcutaneous injection of SVF in the fingers of twelve patients to be proven. Secondary efficacy endpoints evaluated at 2 months (M2) and 6 months (M6) showed an improvement in disability, pain, severity of Raynaud's phenomenon, trophicity, the number of digital ulcers, hand mobility and in the quality of life. These encouraging results have encouraged the investigators to propose a trial which would bear on a higher number of patients and include a control group.

ELIGIBILITY:
Inclusion Criteria:

* Systemic Sclerosis ( limited or diffuse cutaneous shape)
* Men and women of more than 18 years old
* Patients wishing for a therapeutic alternative
* Functional Disability of the dominant hand authenticated by a functional index of the hand of Cochin functional scale upper to 20

Exclusion Criteria:

* Body mass index (weight in kilograms divided by height in meters squared) lower than 18
* Finger infection (including infected ulcer, ulcer with signs of local inflammation and clinical suspicion of osteitis)
* Contraindication to surgery
* Prescription of a new systemic treatment for SSc in the month before the inclusion
* Subjects infected with HIV, HCV ( hepatitis C virus) , HBV (hepatitis B virus), HTLV ( human T-cell leukemia virus) and syphilis
* Pre-menopausal women of reproductive age, taking no contraceptive method
* Patients receiving immunosuppressive therapy not including corticosteroid therapy < 10 mg/D and methotrexate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Cochin hand functional scale | 3 months
  effects of SVF injections in the fingers of patients suffering from SSc evaluated at 3 months, in comparison to the control group

SECONDARY OUTCOMES:
the pain in the hands (EVA pain scale), | 6 months
  effects of SVF injections in the fingers of patients suffering from SSc on evaluated at 1.3 and 6 months, in comparison to the control group
the quality of life- score adapted to scleroderma (SHAQ) | 6 months
  effects of SVF injections in the fingers of patients suffering from SSc , evaluated at 1.3 and 6 months, in comparison to the control group
the mobility(score de Kapandji et distance pulpe/pli palmaire distal) | 6 months
  effects of SVF injections in the fingers of patients suffering from SSc , evaluated at 1.3 and 6 months, in comparison to the control group
the strength(Jamar et Pinch test) | 6 months
  effects of SVF injections in the fingers of patients suffering from SSc , evaluated at 1.3 and 6 months, in comparison to the control group
the finger tactile sensitivity | 6 months
  effects of SVF injections in the fingers of patients suffering from SSc , evaluated at 1.3 and 6 months, in comparison to the control group
the trouble trophicity (health assesment questionnaire) | 6 months
  effects of SVF injections in the fingers of patients suffering from SSc , evaluated at 1.3 and 6 months, in comparison to the control group concerning trophicity: Rodnan score modified for the hand, finger circumference with a ring sizer, monitoring of existing ulcers and of the onset of new ulcers
the severity (frequency and intensity of crises) of Raynaud's phenomenon | 6 months
  effects of SVF injections in the fingers of patients suffering from SSc , evaluated at 1.3 and 6 months, in comparison to the control group concerning severity of Raynaud's phenomenon
the vascular suppression score | 6 months
  effects of SVF injections in the fingers of patients suffering from SSc , evaluated at 1.3 and 6 months, in comparison to the control group concerning vascular suppression score calculated using nail-fold capillaroscopy

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte GRANEL, MD, Principal Investigator — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

REFERENCES:
- [Derived] Daumas A, Magalon J, Jouve E, Casanova D, Philandrianos C, Abellan Lopez M, Mallet S, Veran J, Auquit-Auckbur I, Farge D, Levesque H, Benhamou Y, Arnaud L, Giraudo L, Dumoulin C, Giverne C, Boyer O, Giuliani A, Bourgarel V, Harle JR, Schleinitz N, Brunet J, Pers YM, Ferreira R, Cras A, Boccara D, Larghero J, Chateau J, Hot A, Dignat-George F, Magalon G, Sabatier F, Granel B. Adipose tissue-derived stromal vascular fraction for treating hands of patients with systemic sclerosis: a multicentre randomized trial Autologous AD-SVF versus placebo in systemic sclerosis. Rheumatology (Oxford). 2022 May 5;61(5):1936-1947. doi: 10.1093/rheumatology/keab584. PMID 34297066